CLINICAL TRIAL: NCT07138105
Title: Artificial Intelligence in Surgical Practice in Sudan: Feasibility, Barriers, and Ethical Perspectives From a National Cross-Sectional Survey of Doctors
Brief Title: Artificial Intelligence in Surgical Practice in Sudan: National Survey of Doctors
Acronym: NASAPS
Status: Enrolling by invitation | Type: Observational
Sponsor: Sudan Medical Specialization Board (Other Government)
Responsible Party: Principal Investigator, Alsadig Suliman, Principal Investigator, Sudan Medical Specialization Board
Other Study IDs: MOH-NAT-SURG-AI-2025
Record Dates: First submitted 2025-08-15; First posted 2025-08-22 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Surgical Procedures, Operative; Artificial Intelligence (AI); Wounds and Injuries; War Injury; Health Services Accessibility; Hospitals; Developing Countries
Keywords: Artificial Intelligence; Surgery; Sudan; National Survey; Surgical Practice; Health System Resilience; Conflict Zones; Low-Resource Settings; Triage; Telemedicine; Surgical Education; Offline AI Tools
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: National AI in Surgical Practice Survey - Sudan — An online, cross-sectional national survey targeting Sudanese doctors who provide surgical care in any capacity. The survey collects data on awareness, prior experience, perceived benefits, barriers, and training needs for adopting artificial intelligence in surgical practice. Participants include house officers, medical officers, registrars/residents, specialists, consultants, and general practitioners performing surgical procedures in public, private, NGO, or military hospitals. The study does not involve the implementation or testing of AI tools but aims to inform the design of future AI solutions tailored for low-resource and conflict-affected health systems.

SUMMARY:
This is a national survey of doctors in Sudan who are involved in providing surgical care. The aim is to understand their awareness, experiences, and opinions about using artificial intelligence (AI) in surgery. The survey includes all cadres-house officers, medical officers, registrars, residents, specialists, consultants, and general practitioners who perform surgical procedures-working in public, private, NGO, and military hospitals across Sudan.

Participants are asked about their familiarity with AI, barriers to its use (such as poor infrastructure, lack of training, or cost), interest in training, and possible uses in Sudan's health system, especially in conflict-affected areas. The study does not test any AI tools but collects information to help design future AI solutions that work offline, in low-bandwidth conditions, and meet the needs of surgeons and surgical teams in Sudan.

ELIGIBILITY:
Inclusion Criteria:

* Sudanese doctors currently practicing in Sudan. Provides surgical care in any capacity (house officer/intern, medical officer, registrar/resident, specialist/consultant, general practitioner performing surgical procedures).
* Works in any sector: public, private, NGO, or military hospital/clinic.

Exclusion Criteria:

* Not currently practicing in Sudan.
* Non-clinicians, students without surgical patient care roles.
* Duplicate or incomplete survey responses.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All Sudanese doctors actively providing surgical care across Sudan, including house officers, medical officers, registrars/residents, specialists, consultants, and general practitioners who perform surgical procedures. Participants may work in public, private, NGO, or military facilities, in both rural and urban settings. The population represents a wide range of surgical experience levels and facility types, providing a comprehensive national perspective on artificial intelligence readiness in surgical practice.
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2025-02-01 (Actual); Primary Completion 2025-12-20 (Estimated); Study Completion 2025-12-20 (Estimated)

PRIMARY OUTCOMES:
Awareness of Artificial Intelligence in Surgical Practice Among Doctors in Sudan | At survey completion (Feb 2025 - Dec 2025)
  Percentage of Sudanese doctors providing surgical care who report being aware of artificial intelligence applications in surgical practice. Awareness will be measured using a validated questionnaire adapted from established AI readiness and awareness tools, covering familiarity with AI concepts, knowledge of clinical applications, and perceived relevance to surgical care in Sudan

CONTACTS AND LOCATIONS:
Locations (1):
- Khartoum Teaching Hospital, Khartoum, Khartoum State, Sudan

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared because the dataset contains sensitive information from doctors working in conflict-affected regions of Sudan. Even with anonymization, the small and specialized population could allow re-identification. Only aggregated, de-identified results will be reported publicly.